CLINICAL TRIAL: NCT07247487
Title: Comparative Analysis of Diet and Cardiometabolic Health in Individuals Following Vegan, Vegetarian, and Omnivorous Diets in the City of Rosario
Brief Title: Diet and Cardiometabolism in Rosario
Acronym: DiCaMeR
Status: Recruiting | Type: Observational
Sponsor: Universidad del Centro Educativo Latinoamericano (Other)
Collaborators: Universidad Nacional de Rosario (Other)
Responsible Party: Principal Investigator, Ariel Kraselnik, Medical Doctor, Professor, Universidad del Centro Educativo Latinoamericano
Other Study IDs: NUT 817
Record Dates: First submitted 2025-11-16; First posted 2025-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular (CV) Risk; Nutrition; Cardiometabolic Health Indicators
Keywords: Vegan; Vegetarian; Plant-based; Cardiometabolic health; Cardiometabolism; Cardiovascular health; Diet; Nutrition; Dietary Patterns; Nutrients
MeSH Terms: interventions — Diet, Vegan; Diet, Vegetarian

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vegan: Consumption of meat (including red meat, poultry or fish), dairy products or eggs less than once per month.
  Interventions: Behavioral: Vegan diet
- Vegetarian: Consumption of meat (including red meat, poultry, or fish) less than once per month, with regular consumption of dairy products and/or eggs.
  Interventions: Behavioral: Vegetarian diet
- Omnivorous: Regular consumption of meat (including red meat, poultry or fish), dairy products, and/or eggs.
  Interventions: Behavioral: Omnivorous diet

INTERVENTIONS:
Behavioral: Vegan diet — Individuals reporting consumption of meat (including red meat, poultry, or fish), dairy products, and eggs less than once per month.
  Groups: Vegan
Behavioral: Vegetarian diet — Individuals reporting consumption of meat (including red meat, poultry, or fish) less than once per month, with regular consumption of dairy products and/or eggs.
  Groups: Vegetarian
Behavioral: Omnivorous diet — Individuals reporting regular consumption of meat (including red meat, poultry, or fish), dairy products, and/or eggs.
  Groups: Omnivorous

SUMMARY:
The DiCaMeR study is an observational, cross-sectional study aimed at evaluating the relationship between dietary patterns and cardiometabolic health in adults. The study includes adults following vegan, vegetarian, and omnivorous diets residing in Rosario, Argentina. Participants undergo comprehensive assessments including dietary intake, anthropometric measurements, body composition, blood pressure, grip strenght, and laboratory biomarkers related to cardiovascular and metabolic health. The main objective is to compare diet characteristics and cardiometabolic risk profiles across different dietary patterns, providing insights into the potential health benefits and risks associated with each dietary pattern.

DETAILED DESCRIPTION:
This study will collect demographic, medical, dietary, and biochemical data to evaluate differences among vegan (VGN), ovo-lacto-vegetarian (OLV), and omnivorous (OMNI) participants. Demographic information will include age, sex, district of residence, marital status, number of children, occupation, health coverage (public, social security, or private), and highest educational level attained. Questions were adapted from the Argentine National Surveys of Households and Risk Factors.

Medical history will include current or past significant diseases, psychiatric conditions, reproductive status (premenopausal or menopausal), and habitual medication use. Participants taking drugs that may alter study outcomes (such as antihypertensives, lipid-lowering agents, or oral contraceptives) within the past 6 months will be excluded. Tobacco use will be classified as current, former, or never smoker. Information on supplement use and alcohol intake will also be collected. Alcohol consumption will be categorized as non-drinker, within recommended limits (up to one drink per day for women and two for men), or risk drinker (above these limits). Physical activity will be evaluated using the International Physical Activity Questionnaire (IPAQ) in it's short version, allowing classification into low, moderate, or high activity levels.

Self-perceived quality of life will be assessed with the EQ5D-3L questionnaire validated in Argentina, covering five health dimensions (mobility, self-care, daily activities, pain/discomfort, and anxiety/depression). Following national survey methodology, answers will be grouped into "no problem" or "some problem."

Dietary satisfaction will be evaluated using the DSat-28 questionnaire, which measures satisfaction in domains such as healthy lifestyle, eating out, cost, and food concerns. Higher scores indicate greater satisfaction.

Physical examination will include blood pressure measurement (validated automatic device), weight, height, and waist circumference according to WHO standards. Body composition will be assessed using bioelectrical impedance analysis (BIA), a validated method showing high correlation with DXA. Maximum voluntary isometric grip strength assessed with a calibrated hand dynamometer.

Participants will self-report their dietary pattern as vegan (VGN), ovo-lacto-vegetarian (OLV), or omnivorous (OMNI). They will also indicate the estimated month and year of diet adoption and their main motivation (ethics, environment, health, taste, religion, spirituality, habit, or other). Dietary intake will be recorded for three days (two weekdays and one weekend day), and nutrient composition will be analyzed using MAR24 software, validated for the Argentine population.

Fasting blood samples (12 hours) will be obtained to determine hematological, metabolic, and biochemical parameters. These include complete blood count, renal and liver function (urea, creatinine, AST, ALT, alkaline phosphatase, bilirubin, total proteins, albumin), lipid profile (total, HDL, and LDL cholesterol, triglycerides, apolipoprotein B), glucose and HbA1c, insulin (for HOMA-IR calculation), thyroid function (TSH), inflammation (high-sensitivity C-reactive protein), uric acid, vitamin B12, homocysteine, and iron status (serum iron, transferrin, percentage of transferrin saturation, and ferritin).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Residence in the city of Rosario or surrounding areas.
* Without major diseases.
* BMI >18.5 and <30.
* Adherence to a vegan, vegetarian, or omnivorous diet for at least 1 consecutive year at the time of recruitment.

Exclusion Criteria:

* Acute or chronic diseases (cancer, infections, heart disease, or others), gastrointestinal disorders affecting diet, diabetes mellitus, chronic kidney or liver disease, or any other condition that could affect study outcomes.
* Food allergies or intolerances that substantially affect the individual's usual diet.
* Pregnant or breastfeeding women.
* High-performance athletes (>15 hours per week of high-intensity physical activity).
* Use of medications that could affect study outcomes, including antihypertensives, lipid-lowering drugs, hypoglycemic agents, glucocorticoids, and anti-obesity drugs. Note: vitamin, mineral, or other dietary supplements are not exclusion criteria.
* Problematic use of alcohol or other drugs.
* Simultaneous participation in another clinical trial.
* Inability (physical or psychological) to perform the procedures required by this study.
* Blood transfusions within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-65 years from Rosario, Argentina, following a vegan, vegetarian, or omnivorous diet for ≥1 year. Generally healthy, BMI 18.5-30. Excludes pregnant or breastfeeding women, high-performance athletes, individuals with major diseases, problematic alcohol or drug use, recent blood transfusions, or those unable to complete study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Diet Composition | 12/2025 - 12/2027
  Descriptive and comparative analysis of vegan, vegetarian and omnivorous diets. Dietary intake estimation through validated questionnaires and tools to estimate nutrient composition.
Total Cholesterol | 12/2025 - 12/2027
  Serum total cholesterol concentration (mg/dl)
LDL-Cholesterol | 12/2025 - 12/2027
  Serum LDL cholesterol concentration calculated by Friedewald equation (mg/dl)
HDL-Cholesterol | 12/2025 - 12/2027
  Serum HDL-cholesterol concentration (mg/dl)
Triglycerides | 12/2025 - 12/2027
  Serum triglycerides concentration (mg/dl)
Fasting glucose | 12/2025 - 12/2027
  Serum fasting glucose concentration (mg/dl)
HbA1c | 12/2025 - 12/2027
  Glycated hemoglobin percentage (%)
Fasting Insulin | 12/2025 - 12/2027
  Serum fasting insulin concentration (µIU/mL)
HOMA-IR | 12/2025 - 12/2027
  Homeostatic Model Assessment of Insulin Resistance, calculated using fasting glucose and fasting insulin concentrations.
High-sensitivity C-reactive Protein | 12/2025 - 12/2027
  Serum High-sensitivity C-reactive Protein concentration (mg/L)
Uric Acid | 12/2025 - 12/2027
  Serum uric acid concentration (mg/dL)
Vitamin B12 | 12/2025 - 12/2027
  Serum vitamin B12 concentration (pg/mL)
Homocysteine | 12/2025 - 12/2027
  Plasma homocysteine concentration (µmol/L)
25-hydroxy Vitamin D | 12/2025 - 12/2027
  Serum 25(OH)D concentration (ng/mL)
Serum Iron | 12/2025 - 12/2027
  Serum iron concentration (µg/dL)
Ferritin | 12/2025 - 12/2027
  Serum ferritin concentration(ng/mL)
Transferrin | 12/2025 - 12/2027
  Serum transferrin concentration(mg/dL)
Transferrin Saturation | 12/2025 - 12/2027
  Percentage of transferrin saturation calculated from serum iron and total iron-binding capacity (%)
Complete Blood Count (CBC) | 12/2025 - 12/2027
  Hemoglobin, hematocrit, red blood cell indices (MCV, MCH, MCHC), red blood cell count, white blood cell count (including differential), and platelet count as reported by the laboratory.
Blood Pressure | 12/2025 - 12/2027
  Systolic and diastolic blood pressure measured in mmHg using a validated automated device.
Body Weight | 12/2025 - 12/2027
  Body weight measured in kilograms (kg) using a calibrated scale.
Body Mass Index (BMI) | 12/2025 - 12/2027
  BMI calculated as weight divided by height squared (kg/m²).
Waist Circumference | 12/2025 - 12/2027
  Waist circumference measured in centimeters (cm) at the midpoint between the last rib and the iliac crest.
Hip Circumference | 12/2025 - 12/2027
  Hip circumference measured in centimeters (cm) at the level of the greater trochanters.
Waist-to-Hip Ratio | 12/2025 - 12/2027
  Waist-to-hip ratio calculated as waist circumference divided by hip circumference (unitless).
Body Composition (Fat Mass and Lean Mass) | 12/2025 - 12/2027
  Total body fat mass and lean mass measured using bioelectrical impedance analysis (kg and %).

SECONDARY OUTCOMES:
Supplement use | 12/2025 - 12/2027
  Type, dosing and if it was prescribed by a a health professional.
Satisfaction with the current diet | 12/2025 - 12/2027
  D-Sat 28 Questionnaire
Physical activity levels and global quality of life | 12/2025 - 12/2027
  IPAQ and EQ5D-3L Questionnaires
Reasons for adopting dietary patterns | 12/2025 - 12/2027
  Ethics / animal rights, Environment, Health, Taste, Religion/Spirituality, Custom, Other (specify)
Alcohol and tobacco use | 12/2025 - 12/2027
Serum Urea | 12/2025 - 12/2027
  Serum urea concentration (mg/dL).
Serum Creatinine | 12/2025 - 12/2027
  Serum creatinine concentration (mg/dL).
Alanine Aminotransferase (ALT/GPT) | 12/2025 - 12/2027
  Serum alanine aminotransferase concentration (U/L).
Aspartate Aminotransferase (AST/GOT) | 12/2025 - 12/2027
  Serum aspartate aminotransferase concentration (U/L).
Alkaline Phosphatase (ALP) | 12/2025 - 12/2027
  Serum alkaline phosphatase concentration (U/L).
Bilirubin | 12/2025 - 12/2027
  Serum total bilirubin concentration (mg/dL).
Bilirubin | 12/2025 - 12/2027
  Serum total and direct bilirubin concentration (mg/dL).
Total Protein | 12/2025 - 12/2027
  Serum total protein concentration (g/dL).
Thyroid-Stimulating Hormone (TSH) | 12/2025 - 12/2027
  Serum thyroid-stimulating hormone concentration (µIU/mL).
Grip Strength | 12/2025 - 12/2027
  Maximum voluntary isometric grip strength assessed with a calibrated hand dynamometer. The recorded value is the highest (kg) obtained from three valid attempts using the participant's dominant hand.

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Consultorios Prisma, Rosario, Santa Fe Province
  - Universidad del Centro Educativo Latinoamericano, Rosario, Santa Fe Province

IPD SHARING:
Plan to Share IPD: Undecided
Data available under request for research purposes, and after evaluation by the investigators.

REFERENCES:
- See also: Official study website — https://nutricionbasadaenplantas.com/page/dicamer